CLINICAL TRIAL: NCT06631833
Title: The Effects of Psychosocial Factors in Physical Activity Promotion Among Overweight and Obese Children in Yunnan Province, China Using Youth Physical Activity Promotion Model
Brief Title: Effects of an Adolescent Physical Activity Promotion Model on Physical Activity in Obese Chinese Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Han Mingxue, Dr., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USM/JEPeM/KK/23010097
Record Dates: First submitted 2024-09-28; First posted 2024-10-08 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Obesity Prevention
Keywords: Overweight and obese children; physical activity
MeSH Terms: conditions — Overweight; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group 48 persons(YPAP) (Experimental): Intervention measures based on the YPAP model.
  Interventions: Behavioral: Intervention measures based on the YPAP model.
- Control group 48 persons (No Intervention): No intervention was used in the control group.

INTERVENTIONS:
Behavioral: Intervention measures based on the YPAP model. — The intervention group received an 8-week intervention program aimed at gradually increasing their physical activity levels. The intervention program included the following components: 1) 1-2 sessions of moderate-intensity physical activity per week, each lasting 45 minutes, with activities provided by physical activity experts; 2) one health education lecture every two weeks, each lasting 60 minutes; and 3) one family physical activity session per week, each lasting 30 minutes at a lower intensity. At the end of the intervention period, relevant questionnaires were used for measurement.
  Arms: Intervention group 48 persons(YPAP)

SUMMARY:
The purpose of this study was to evaluate the effectiveness of an intervention program based on the Youth Physical Activity Promotion Model (YPAP) in increasing physical activity levels among overweight and obese children in China.

DETAILED DESCRIPTION:
This observational study aims to understand the impact of a YPAP-based intervention on the psychosocial factors and physical activity of overweight and obese children aged 12-15 in China. The intervention consists of three key components: 1) The intervention group received an 8-week intervention program aimed at gradually increasing their physical activity levels. The intervention program included the following components: 1) 1-2 sessions of moderate-intensity physical activity per week, each lasting 45 minutes, with activities provided by physical activity experts; 2) one health education lecture every two weeks, each lasting 60 minutes; and 3) one family physical activity session per week, each lasting 30 minutes at a lower intensity. At the end of the intervention period, relevant questionnaires were used for measurement.

ELIGIBILITY:
Inclusion Criteria:

* Chinese children
* Aged between 12 and 15 years
* Able to complete questionnaires before and after the intervention
* Children who meet the standards for overweight and obesity among Chinese school-age children

Exclusion Criteria:

* Children with serious health issues (e.g., heart disease, respiratory diseases, severe musculoskeletal disorders) or those advised by a doctor not to participate in physical activities.
* Children currently involved in other intervention programs that affect physical activity or weight.
* Children without written consent from their parents or guardians.
* Children on long-term medication that might affect physical activity or weight (as determined by parents and teachers).

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
The Youth Physical Activity Promotion Model (YPAP) was used to assess changes in physical activity (PA) among overweight and obese children in Yunnan Province, China. | 12 weeks
  The study measured the total physical activity of the control and experimental groups before and after the intervention (pre-test and post-test). The Physical Activity Questionnaire for Adolescents (PAQ-A) was used for self-reported measurements, calculating changes in PAQ-A scores before and after the intervention. Repeated measures ANOVA was applied to evaluate the effects of time, group, and their interaction, with significance set at p < 0.05, and effect sizes reported using partial eta-squared (η²).
The Youth Physical Activity Promotion Model (YPAP) was used to assess changes in self-efficacy among overweight and obese children in Yunnan Province, China. | 12 weeks
  The study measured the changes in self-efficacy of the control and experimental groups before and after the intervention (pre-test and post-test) using the General Self-Efficacy Scale (GSES), which employs a 5-point Likert scale. Researchers calculated the changes in GSES scores for both groups. Repeated measures ANOVA was used to evaluate the effects of time, group, and their interaction, with significance set at p < 0.05, and effect sizes reported using partial eta-squared (η²).
The Youth Physical Activity Promotion Model (YPAP) was used to assess changes in enjoyment of physical activity among overweight and obese children in Yunnan Province, China. | 12 weeks
  The study measured the changes in enjoyment levels of the control and experimental groups before and after the intervention (pre-test and post-test) using the Physical Activity Enjoyment Scale (PACES), which employs a 5-point Likert scale. Researchers calculated the changes in PACES scores for both groups. Repeated measures ANOVA was used to evaluate the effects of time, group, and their interaction, with significance set at p < 0.05, and effect sizes reported using partial eta-squared (η²).
he Youth Physical Activity Promotion Model (YPAP) was used to assess changes in perceived competence among overweight and obese children in Yunnan Province, China. | 12 weeks
  The study measured changes in perceived competence of the control and experimental groups before and after the intervention (pre-test and post-test) using the Children's Physical Activity Correlates Scale (CPAC-C), which employs a 4-point Likert scale. Researchers calculated the changes in CPAC-C scores for both groups. Repeated measures ANOVA was applied to evaluate the effects of time, group, and their interaction, with significance set at p < 0.05, and effect sizes reported using partial eta-squared (η²).

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Hairul Anuar Hashim, Dr, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Zhaotong Junior Middle School, Yunnan Province, China, Zhaotong, Yunnan, China

IPD SHARING:
Plan to Share IPD: No